CLINICAL TRIAL: NCT03931161
Title: Effect of Evolocumab on Carotid Plaque Composition in Asymptomatic Carotid Artery Stenosis
Brief Title: Effect of Evolocumab on Carotid Plaque Composition in Asymptomatic Carotid Artery Stenosis (EVOCAR-1)
Acronym: EVOCAR-1
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Imperial College Healthcare NHS Trust (Other)
Collaborators: Imperial College London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EVOCAR-1
Record Dates: First submitted 2019-04-15; First posted 2019-04-30 (Actual); Last update posted 2022-10-13 (Actual); Status verified 2022-10

CONDITIONS: Carotid Artery Stenosis
Keywords: carotid plaque morphology; carotid plaque composition; evolocumab
MeSH Terms: conditions — Carotid Stenosis | interventions — evolocumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo (Placebo Comparator): Matching Placebo.
  Interventions: Drug: Placebo Auto-Injector
- Evolocumab (Active Comparator): Evolocumab Auto-Injector [Repatha]
  Interventions: Drug: Evolocumab Auto-Injector [Repatha]

INTERVENTIONS:
Drug: Evolocumab Auto-Injector [Repatha] — Auto-Injector, 140 mg every two weeks.
  Other Names: Repatha
  Arms: Evolocumab
Drug: Placebo Auto-Injector — Matching Placebo for the active comparator (Evolocumab)
  Other Names: Placebo
  Arms: Placebo

SUMMARY:
This is a phase IV, randomised, placebo-controlled, double-blind, parallel group study to determine the effect of Evolocumab treatment on carotid plaque morphology and composition in asymptomatic patients with >50% carotid artery stenosis.

DETAILED DESCRIPTION:
In this study patients will be randomised in a 1:1 ratio to receive Evolocumab 140 mg every two weeks or matching placebo, to be administered for 12 months. After 12 months of treatment, patients will remain in follow-up for a further 12 months.

High resolution magnetic resonance imaging (MRI) will be used to serially monitor the impact of Evolocumab on carotid plaque morphology and composition in patients with significant carotid stenosis who do not meet clinical criteria for carotid endarterectomy. This approach will reveal if clinically beneficial plaque regression occurs, without requiring the large patient cohorts or long follow-up needed for cardiovascular outcome trials.

Results from this study will establish whether treatment with Evolocumab is likely to be beneficial to patients with asymptomatic carotid stenosis.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Sufficient English language ability to adequately understand the study
* Able to give informed consent
* Significant carotid artery plaque with 50-70% stenosis on ultrasound or MRI performed prior to screening
* Significant asymptomatic carotid artery plaque with >70% stenosis on ultrasound or MRI performed prior to screening, but carotid endarterectomy or carotid artery stenting has been deemed unsuitable by multidisciplinary team during routine clinical care
* Lipid-rich necrotic core (LRNC) on baseline MRI scan
* Adequate image quality for MRI analysis.
* LDL-C ≥2.6 mmol/L (100 mg/dL)
* On stable dose of maximally-tolerated lipid-lowering therapy in accordance with UK national clinical guidelines (NICE CG18120) for ≥2 months prior to screening. Acceptable non-statin lipid-lowering medications include ezetimibe or a fibrate.

Exclusion Criteria:

* Any medical condition which, in the opinion of the investigators, would present an unacceptable risk to the participant if they were to take part in the trial, or prevent them from following the trial protocol
* Current or previous treatment with a PCSK9 inhibitor
* Eligible for PCSK9 inhibitor treatment under current NICE guidelines
* Contra-indication to or inability to use Evolocumab treatment, including:

  * Sensitivity to Evolocumab or any associated excipients
  * Unable to tolerate or perform self-administration of Evolocumab by auto-injector
  * Lack of suitable refrigerated storage
* Contra-indication to or inability to tolerate MRI
* Estimated glomerular filtration rate (eGFR) ≤45 mL/min/1.73 m2 prior to MRI scan
* Pregnancy or breast-feeding
* Women of childbearing potential who are unwilling or unable to use a highly effective method of contraception

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2019-09-04 (Actual); Primary Completion 2023-05-06 (Estimated); Study Completion 2024-05-06 (Estimated)

PRIMARY OUTCOMES:
Change in lipid-rich necrotic core | 12 months
  Change in lipid-rich necrotic core (LRNC) size at 12 months, compared to baseline

SECONDARY OUTCOMES:
Percentage of LRNC core | 12 months
  Change in percentage lipid-rich necrotic core (LRNC) at 12 months, compared to baseline
LRNC regression | 12 months
  Percentage of participants achieving LRNC regression at 12 months
LRNC volume | 24 months
  Change in carotid plaque LRNC volume at other time-points, compared to baseline
LRNC percentage | 24 months
  Change in carotid plaque LRNC percentage at other time-points, compared to baseline
Measures of other carotid plaque burden - Volume wall thickness | 24 months
  Absolute and percentage change, compared to baseline, of volume wall thickness
Measures of other carotid plaque burden - Volume wall area | 24 months
  Absolute and percentage change, compared to baseline, volume wall area
Measures of other carotid plaque burden - Calcification | 24 months
  Absolute and percentage change, compared to baseline, of plaque composition (calcification)
Measures of other carotid plaque burden - Fibrous tissue volume | 24 months
  Absolute and percentage change, compared to baseline, of plaque composition (fibrous tissue volume)
Measures of other carotid plaque burden - New intra-plaque haemorrhage | 24 months
  Absolute and percentage change, compared to baseline, of plaque composition (new intra-plaque haemorrhage)

OTHER OUTCOMES:
Exploratory outcomes 1: Change in biochemical parameters - total cholesterol | 24 months
  Absolute and percentage change compared to baseline in total cholesterol.
Exploratory outcomes 1: Change in biochemical parameters - LDL-C | 24 months
  Absolute and percentage change compared to baseline in LDL-C.
Exploratory outcomes 1: Change in biochemical parameters - HDL-C | 24 months
  Absolute and percentage change compared to baseline in high density lipoprotein-associated cholesterol (HDL-C).
Exploratory outcomes 1: Change in biochemical parameters - triglycerides | 24 months
  Absolute and percentage change compared to baseline in triglycerides.
Exploratory outcomes 1: Change in biochemical parameters - lipoprotein (a) | 24 months
  Absolute and percentage change compared to baseline in lipoprotein(a).
Exploratory outcomes 2: Number of patients with Cardio & cerebrovascular events - Ischaemic and non-ischaemic stroke | 24 months
  Cardio- and cerebrovascular events [be adjudicated by the Investigators], including: Ischaemic and non-ischaemic stroke
Exploratory outcomes 2: Number of patients with Cardio & cerebrovascular events - TIA | 24 months
  Cardio- and cerebrovascular events [be adjudicated by the Investigators], including: Transient ischaemic attack
Exploratory outcomes 2: Number of patients with Cardio & cerebrovascular events - Progression to carotid endarterectomy | 24 months
  Cardio- and cerebrovascular events [be adjudicated by the Investigators], including: Progression to carotid endarterectomy
Exploratory outcomes 2: Number of patients with Cardio & cerebrovascular events - MI | 24 months
  Cardio- and cerebrovascular events [be adjudicated by the Investigators], including: Myocardial infarction
Exploratory outcomes 2: Number of patients with Cardio & cerebrovascular events - Unstable angina | 24 months
  Cardio- and cerebrovascular events [be adjudicated by the Investigators], including: Unstable angina
Exploratory outcomes 2: Number of patients with Cardio & cerebrovascular events - Hospitalisation for heart failure | 24 months
  Cardio- and cerebrovascular events [be adjudicated by the Investigators], including: Hospitalisation for heart failure
Exploratory outcomes 2: Number of patients with Cardio & cerebrovascular events -PAD-related end points: peripheral revascularization, | 24 months
  Cardio- and cerebrovascular events [be adjudicated by the Investigators], including: PAD-related end points: peripheral revascularization,

CONTACTS AND LOCATIONS:
Overall Officials: Jaimini Cegla, BSc MSc MBBS MRCP FRCPath PhD, Principal Investigator — Imperial College London
Locations (1):
- Imperial College Healthcare NHS Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No